CLINICAL TRIAL: NCT06818929
Title: Relationship Between Active Flexibility and Hamstring Concentric to Eccentric Peak Torque Ratio in Athletes: a Cross-Sectional Study
Brief Title: Relationship Between Active Flexibility and Hamstring Concentric to Eccentric Peak Torque Ratio in Athletes
Acronym: Q/H
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, El.saieed Ahmed Attia, demonstrator, faculty of physical therapy, basic science department, Cairo University
Other Study IDs: P.T.REC/012/005295
Record Dates: First submitted 2025-01-16; First posted 2025-02-11 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Sports Physical Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study measures flexibility using 2D video analysis during the H-test and assesses concentric/eccentric peak torque ratios (H/Q ratio) to determine their importance in returning to sport after a hamstring strain.

DETAILED DESCRIPTION:
This observational cross-sectional study aimed to assess the H:Q peak torque ratio, hamstring Ecc/Con peak torque ratio, and hamstring flexibility during the H-test using 2D video analysis in professional soccer players.

Participants:

Forty-seven participants (mean age: 28 ± 7 years; BMI: 22.98 ± 1.16 kg/m²) were recruited.

Inclusion criteria: History of hamstring strain for more than three months. Exclusion criteria: Recent hamstring injury within the last 3 months, ACL injury within the past 12 months (hamstring graft), lumbar disc issues (L3-L4, L5-S1), or sacroiliac dysfunction.

Sample Size Calculation:

Conducted using G*Power software (version 3.0.10) for a biserial correlation model with a power of 0.80, alpha level of 0.05, and effect size of 0.38.

Minimum of 47 participants, with 10% added for potential dropouts, yielding a total sample size of 52.

Standardization Procedures:

The principal investigator was responsible for all aspects of experimental preparation, including providing instructions, adjusting the isokinetic machine, attaching adaptors, placing braces, identifying bony landmarks, and collecting data.

The chair, dynamometer, and adaptor settings were configured according to CSMI guidelines to enhance inter-rater reliability.

Participants received standardized instructions on the warm-up process, isokinetic testing, and performing the H-test.

Familiarization sessions for both the isokinetic and H-tests were conducted beforehand using submaximal effort to ensure participants were well-versed in the procedures.

H-test:

The primary outcome measure, hamstring active flexibility, was assessed by measuring the range of motion during hip flexion.

Participants were positioned supine on a table with straps securing the contralateral leg, hip, and trunk to ensure stability and correct posture throughout the test.

Two visual markers were placed on the greater trochanter and lateral malleolus of the tested limb.

A knee support (Orthopedic Bracewear Air-X©) was applied to the tested limb to maintain knee extension and prevent flexion during the movement.

The procedure began with a warm-up consisting of three slow hip flexions, followed by three maximum-velocity trials, each separated by 5 seconds of rest.

Hip flexion was recorded using a smartphone (iPhone 12©, 30 Hz) mounted on a tripod positioned 3 meters from the participant and 1 meter in height.

Participants performed hip flexions at maximum speed and ROM while maintaining full knee extension.

The angle between the visual markers was captured through 2D video recording during each trial.

The recorded video footage was analyzed using Kinovea software (version 0.9.5) to calculate the hip flexion ROM.

Peak Torque Ratios Assessment:

The Cybex Norm isokinetic dynamometer was utilized for measurements of hamstring Ecc/Con peak torque as well as H:Q ratio.

Participants began with a 5-minute warm-up on a stationary bike, followed by dynamic stretching exercises.

For the hamstring Ecc/Con ratio assessment, participants were positioned prone on the isokinetic dynamometer with the knee axis aligned with the dynamometer's axis of rotation.

Familiarization sets consisting of submaximal-effort repetitions were performed.

Maximal-effort repetitions were conducted, and the highest peak torque achieved during eccentric and concentric contractions was recorded.

The Ecc/Con ratio was calculated by dividing the peak torque from eccentric contractions by the peak torque from concentric contractions.

For the H:Q ratio test, participants were seated on the isokinetic dynamometer with the knee axis aligned with the dynamometer's axis of rotation.

Familiarization sets were performed, followed by maximal-effort repetitions to assess the peak torque produced by both the hamstrings and quadriceps.

The H:Q ratio was calculated by dividing the peak torque of the hamstrings by that of the quadriceps.

Data Processing and Statistical Analysis:

Data were analyzed using Python (version 3.10). Descriptive statistics summarized participant characteristics and outcomes. Normality of data was confirmed using the Shapiro-Wilk test. Pearson correlation was applied to examine relationships between H-test scores, Ecc/Con ratio, and H:Q ratio.

Multiple regression analyses assessed the influence of H-test scores and age on torque ratios, including interaction terms for combined effects.

Subgroup analyses stratified participants into age groups (≤25 years and >25 years) to explore age-related differences, with significance set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Football players registered in the Egyptian Football Association.
* Football players with a history of hamstring strain for more than three months.

Exclusion Criteria:

* Hamstring strain less than three months.
* ACL injury within the past 12 months (hamstring graft).
* Lumbar disc issues (L3-L4, L5-S1).
* Sacroiliac pain or dysfunction.

Ages: 21 Years to 34 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: - Male football players registered in the Egyptian Football Association with a history of hamstring strain for more than three months from Egyptian Clubs
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Hamstring Active Flexibility | immediately after the procedure
  measuring the range of motion during hip flexion
Peak torque ratios assessment of hamstring | immediately after the procedure
  hamstring Ecc/Con ratio assessment
Peak torque ratios assessment of hamstring to quadriceps | immediately after the procedure
  The H:Q ratio was calculated by dividing the peak torque of the hamstrings by that of the quadriceps

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Ahmed Zayat - Between the Chateaux, Egypt

IPD SHARING:
Plan to Share IPD: Undecided